CLINICAL TRIAL: NCT00071812
Title: A Phase 2, Multi-Center, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Safety, Tolerability, and Efficacy of LymphoStat-B™ Antibody (Monoclonal Anti-BLyS Antibody) in Subjects With Rheumatoid Arthritis (RA)
Brief Title: A Safety and Efficacy Study of LymphoStat-B™ (Monoclonal Anti-BLyS Antibody) in Subjects With Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Human Genome Sciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LBRA01
Record Dates: First submitted 2003-10-31; First posted 2003-11-05 (Estimated); Results first posted 2012-06-25 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Arthritis, Rheumatoid
Keywords: RA
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — belimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo plus SOC (Placebo Comparator)
  Interventions: Drug: Placebo
- Belimumab 1 mg/kg plus SOC (Experimental)
  Interventions: Drug: Belimumab 1 mg/kg
- Belimumab 4 mg/kg plus SOC (Experimental)
  Interventions: Drug: Belimumab 4 mg/kg
- Belimumab 10 mg/kg plus SOC (Experimental)
  Interventions: Drug: Belimumab 10 mg/kg

INTERVENTIONS:
Drug: Placebo — Placebo IV plus standard therapy (SOC) for RA; placebo administered on Days 0, 14, 28, and every 28 days thereafter through 24 weeks in the double-blind period. In the open-label extension period, placebo patients who opted to participate received belimumab 10 mg/kg IV plus SOC every 28 days for an additional 24 weeks.
  Arms: Placebo plus SOC
Drug: Belimumab 1 mg/kg — Belimumab 1 mg/kg IV plus standard therapy (SOC) for RA; belimumab 1 mg/kg administered on Days 0, 14, 28, and every 28 days thereafter through 24 weeks in the double-blind period. In the open-label extension period, patients who opted to participate either continued on the same dose of belimumab or may have been switched to belimumab 10 mg/kg at the investigator's discretion for an additional 24 weeks.
  Other Names: LymphoStat-B®; BENLYSTA®
  Arms: Belimumab 1 mg/kg plus SOC
Drug: Belimumab 4 mg/kg — Belimumab 4 mg/kg IV plus standard therapy (SOC) for RA; belimumab 4 mg/kg administered on Days 0, 14, 28, and every 28 days thereafter through 24 weeks in the double-blind period. In the open-label extension period, patients who opted to participate either continued on the same dose of belimumab or may have been switched to belimumab 10 mg/kg at the investigator's discretion for an additional 24 weeks.
  Other Names: LymphoStat-B®; BENLYSTA®
  Arms: Belimumab 4 mg/kg plus SOC
Drug: Belimumab 10 mg/kg — Belimumab 10 mg/kg IV plus standard therapy (SOC) for RA; belimumab 10 mg/kg administered on Days 0, 14, 28, and every 28 days thereafter through 24 weeks in the double-blind period. In the open-label extension period, patients who opted to participate continued on the same dose of belimumab (10 mg/kg) for an additional 24 weeks.
  Other Names: LymphoStat-B®; BENLYSTA®
  Arms: Belimumab 10 mg/kg plus SOC

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of 3 different doses of belimumab, administered in addition to standard therapy, in patients with rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and efficacy of three different doses of belimumab (1 mg/kg, 4 mg/kg, and 10 mg/kg), administered in addition to standard therapy, compared to placebo plus standard therapy in patients with RA. All patients were to be dosed on Days 0, 14, and 28, then every 28 days for the remainder of 24 weeks. Patients completing the 24-week period could enter a 24-week open-label extension; belimumab patients received the same dose or were switched to 10 mg/kg at the investigator's discretion and former placebo patients received belimumab 10 mg/kg.

ELIGIBILITY:
Primary Inclusion Criteria:

* Diagnosis of RA for at least 1 year
* Failed at least 1 disease modifying anti-rheumatic drug (DMARD) due to toxicity or lack of efficacy. These drugs must include 1 or more of the following: methotrexate, parenteral gold, sulfasalazine, leflunomide, and tumor necrosis factor-alpha (TNFα) inhibitors (infliximab, etanercept or adalimumab)
* Active RA disease of at least moderate disease activity
* Be on a stable RA treatment regimen for at least the past 60 days (for DMARDS); if on non-steroidal anti-inflammatory drugs (NSAIDs) or steroids these must be at a stable dose for the last 30 days

Primary Exclusion Criteria:

* Received a non-FDA approved investigational agent within the last 28 days
* Currently receiving or received within the last 60 days the following: TNFα-inhibitors (infliximab, etanercept, adalimumab) or interleukin-1 receptor antagonist (anakinra)
* Currently receiving or received within the last 6 months the following: anti-CD20 antibody (rituximab) or cyclophosphamide
* Steroid injection into any joint within the last 30 days
* History of hypogammaglobulinemia or immunoglobulin A (IgA) deficiency
* History of chronic infection that has been active within last 6 months, or herpes zoster within last 90 days, or any infection requiring hospitalization or intravenous medication within last 60 days
* Human immunodeficiency virus (HIV), Hepatitis-B, Hepatitis-C

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2003-12; Primary Completion 2005-01 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (63):
- United States (63):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Arthritis Research, Paradise Valley, Arizona
  - University of Arizona, Tucson, Arizona
  - Scripps Clinic, La Jolla, California
  - University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Wallace Rheumatic Disease Center, Los Angeles, California
  - Stanford University School of Medicine, Palo Alto, California
  - Boling Clinical Trials, Rancho Cucamonga, California
  - UCDMC, Sacramento, California
  - Arthritis Care Center, Inc., San Jose, California
  - Arthritis Associates & Osteoporosis Center Of Colorado Springs, Colorado Springs, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Arthritis and Rheumatic Disease Specialties, Aventura, Florida
  - Rheumatology Associates of Central Florida, Orlando, Florida
  - Tampa Medical Group, P.A., Tampa, Florida
  - Radiant Research Boise, Boise, Idaho
  - Institute of Arthritis and Research, Idaho Falls, Idaho
  - Northwestern University Medical School, Chicago, Illinois
  - Rheumatology Associates, Chicago, Illinois
  - Rockford Clinic, Rockford, Illinois
  - Medical Specialists, Munster, Indiana
  - Kentuckiana Center for Better Bone and Joint Health, Louisville, Kentucky
  - Ochsner Clinic Foundation, Baton Rouge, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - The Osteoporosis and Arthritis Clinical Trial Center, Cumberland, Maryland
  - Center for Rhematology and Bone Research, Wheaton, Maryland
  - Tufts - New England Medical Center, Boston, Massachusetts
  - The University of Michigan Health System, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - Arthritis Center of Nebraska, Lincoln, Nebraska
  - Arthritis and Osteoporosis Center, Concord, New Hampshire
  - Strafford Medical Associates, P.A., Dover, New Hampshire
  - The Center For Rheumatology, Albany, New York
  - SUNY-Downstate Medical Center, Brooklyn, New York
  - North Shore University Hospital, Manhasset, New York
  - Jacobi Medical Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Arthritis Clinic and Carolina Bone and Joint, Charlotte, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Stat Research, Inc., Dayton, Ohio
  - McBride Clinic, Oklahoma City, Oklahoma
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Oklahoma Center For Arthritis Therapy & Research, Tulsa, Oklahoma
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh School of Medicine & ASPH, Pittsburgh, Pennsylvania
  - Rheumatic Disease Associates, Willow Grove, Pennsylvania
  - Arthritis Centers of Texas, Dallas, Texas
  - Research Associates of North Texas, Dallas, Texas
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - Houston Institute for Clinical Research, Houston, Texas
  - Texas Research Center, Sugar Land, Texas
  - Arthritis and Rheumatic Diseases Clinic, Morgan, Utah
  - Arthritis Clinic of Northern Virginia, P.C., Arlington, Virginia
  - Edmonds Rheumatology Associates, Edmonds, Washington
  - Evergreen Clinical Reserach, Edmonds, Washington
  - Arthritis Northwest Rheumatology, Spokane, Washington
  - Rheumatology Northwest Clinical Trials, Yakima, Washington
  - Rheumatic Disease Center, Glendale, Wisconsin
  - Gundersen Clinic, Ltd., La Crosse, Wisconsin
  - The Medical College of Wisconsin , Inc, Milwaukee, Wisconsin
  - Marshfield Medical Research Foundation, Wausau, Wisconsin

REFERENCES:
- [Derived] Stohl W, Merrill JT, McKay JD, Lisse JR, Zhong ZJ, Freimuth WW, Genovese MC. Efficacy and safety of belimumab in patients with rheumatoid arthritis: a phase II, randomized, double-blind, placebo-controlled, dose-ranging Study. J Rheumatol. 2013 May;40(5):579-89. doi: 10.3899/jrheum.120886. Epub 2013 Apr 1. PMID 23547209

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Plus SOC: Placebo IV plus standard therapy (SOC) for RA for 24-week double-blind period of the study.
- Belimumab 1 mg/kg Plus SOC: Belimumab 1 mg/kg IV plus standard therapy (SOC) for RA for 24-week double-blind period of the study. The 24-week open-label extension period of the study included patients who completed the 24-week double-blind period and opted to continue to receive the same dose in the 24-week open-label extension period of the study.
- Belimumab 4 mg/kg Plus SOC: Belimumab 4 mg/kg IV plus standard therapy (SOC) for RA for 24-week double-blind period of the study. The 24-week open-label extension period of the study included patients who completed the 24-week double-blind period and opted to continue to receive the same dose in the 24-week open-label extension period of the study.
- Belimumab 10 mg/kg Plus SOC: Belimumab 10 mg/kg IV plus standard therapy (SOC) for RA for 24-week double-blind period of the study. The 24 week-open label extension period of the study included patients who completed the 24-week double-blind period and opted to continue in the 24-week open-label period of the study and included patients who were originally randomized to the belimumab 10 mg/kg group in the double-blind period, patients who switched to belimumab 10 mg/kg at the investigator's discretion, and former placebo patients.
Period: 24-Week Double-Blind Period
Arm/Group | Placebo Plus SOC | Belimumab 1 mg/kg Plus SOC | Belimumab 4 mg/kg Plus SOC | Belimumab 10 mg/kg Plus SOC
Started | 69 | 72 | 71 | 71
Completed | 59 | 66 | 63 | 60
Not Completed | 10 | 6 | 8 | 11
Not completed — Adverse Event | 2 | 3 | 4 | 4
Not completed — Lack of Efficacy | 3 | 1 | 2 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 5 | 1 | 1 | 5
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Period: 24-Week Open-Label Extension Period
Arm/Group | Placebo Plus SOC | Belimumab 1 mg/kg Plus SOC | Belimumab 4 mg/kg Plus SOC | Belimumab 10 mg/kg Plus SOC
Started | 0 (Of 59: 56 switched to 10 mg/kg; 3 elected not to continue in the open-label extension.) | 11 (Of 66: 53 switched to 10 mg/kg; 2 elected not continue in the open-label extension.) | 8 (Of 63: 53 switched to 10 mg/kg; 2 elected not continue in the open-label extension.) | 218 (Of 60: 56 continued with 10 mg/kg; 4 elected not to continue in the open-label extension.)
Completed | 0 | 11 | 7 | 178
Not Completed | 0 | 0 | 1 | 40
Not completed — Adverse Event | 0 | 0 | 0 | 7
Not completed — Lack of Efficacy | 0 | 0 | 0 | 17
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 12
Not completed — Lack of Compliance | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Belimumab 1 mg/kg Plus SOC: Belimumab 1 mg/kg IV plus standard therapy (SOC) for RA for 24-week double-blind period of the study
- Belimumab 4 mg/kg Plus SOC: Belimumab 4 mg/kg IV plus standard therapy (SOC) for RA for 24-week double-blind period of the study
- Belimumab 10 mg/kg Plus SOC: Belimumab 10 mg/kg IV plus standard therapy (SOC) for RA for 24-week double-blind period of the study
- Total: Total of all reporting groups
Arm/Group | Placebo Plus SOC | Belimumab 1 mg/kg Plus SOC | Belimumab 4 mg/kg Plus SOC | Belimumab 10 mg/kg Plus SOC | Total
Number analyzed (Participants) | 69 | 72 | 71 | 71 | 283
Age Continuous [Mean (Standard Deviation); unit: years] | 50.7 (8.8) | 50.6 (8.3) | 50.7 (10.2) | 49.5 (9.3) | 50.4 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 56 | 60 | 54 | 226
  Male | 13 | 16 | 11 | 17 | 57
Region of Enrollment [Number; unit: participants]
  United States | 55 | 61 | 59 | 59 | 234
  Poland | 14 | 11 | 12 | 12 | 49

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With ACR20 (American College of Rheumatology) Response at Week 24, Based on Erythrocyte Sedimentation Rate (ESR)
Description: An ACR20 response is defined as having at least a 20% improvement in tender and swollen joints as well as a 20% improvement in 3 of 5 other criteria (patient assessment, physician assessment, pain scale, disability/functional questionnaire, and acute phase reactant value based on erythrocyte sedimentation rate [ESR]).
Time Frame: Baseline, 24 weeks
Population: Analysis was performed on a modified intention-to-treat (MITT) population, defined as all patients who were randomized and received at least 1 dose of study agent.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Plus SOC | Belimumab 1 mg/kg Plus SOC | Belimumab 4 mg/kg Plus SOC | Belimumab 10 mg/kg Plus SOC
Number analyzed (Participants) | 69 | 72 | 71 | 71
percentage of participants | 15.9 | 34.7 | 25.4 | 28.2
Statistical Analysis 1: Comparison: Placebo Plus SOC vs Belimumab 1 mg/kg Plus SOC; Patients who required rescue RA medications were declared nonresponders, as were patients who dropped out or were missing Week 24 data; Test type: Superiority or Other; p = 0.0097, Likelihood ratio chi-squared — P-value was not adjusted for multiple testing; percent difference from placebo = 18.8, 95% CI 2-sided [4.8 to 32.8]
Statistical Analysis 2: Comparison: Placebo Plus SOC vs Belimumab 4 mg/kg Plus SOC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1677, Likelihood ratio chi-squared — P-value was not adjusted for multiple testing; percent difference from placebo = 9.4, 95% CI 2-sided [-3.9 to 22.7]
Statistical Analysis 3: Comparison: Placebo Plus SOC vs Belimumab 10 mg/kg Plus SOC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0796, Likelihood ratio chi-squared — P-value was not adjusted for multiple testing; percent difference from placebo = 12.2, 95% CI 2-sided [-1.3 to 25.8]

2. Secondary Outcome: Percentage of Patients With an ACR50 Response at Week 24, Based on ESR
Description: An ACR50 response is defined as having at least a 50% improvement in tender and swollen joints as well as a 50% improvement in 3 of 5 other criteria (patient assessment, physician assessment, pain scale, disability/functional questionnaire, and acute phase reactant value based on erythrocyte sedimentation rate [ESR]).
Time Frame: Baseline, 24 weeks
Population: Analysis was performed on a MITT population, defined as all patients who were randomized and received at least 1 dose of study agent.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Plus SOC | Belimumab 1 mg/kg Plus SOC | Belimumab 4 mg/kg Plus SOC | Belimumab 10 mg/kg Plus SOC
Number analyzed (Participants) | 69 | 72 | 71 | 71
percentage of participants | 4.3 | 9.7 | 8.5 | 14.1
Statistical Analysis 1: Comparison: Placebo Plus SOC vs Belimumab 1 mg/kg Plus SOC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2074, Likelihood ratio chi-squared — P-value was not adjusted for multiple testing; percent difference from placebo = 5.4, 95% CI 2-sided [-3.0 to 13.7]
Statistical Analysis 2: Comparison: Placebo Plus SOC vs Belimumab 4 mg/kg Plus SOC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3177, Likelihood ratio chi-squared — P-value was not adjusted for multiple testing; percent difference from placebo = 4.1, 95% CI 2-sided [-4.0 to 12.2]
Statistical Analysis 3: Comparison: Placebo Plus SOC vs Belimumab 10 mg/kg Plus SOC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0418, Likelihood ratio chi-squared — P-value was not adjusted for multiple testing; percent difference from placebo = 9.7, 95% CI 2-sided [0.3 to 19.2]

3. Secondary Outcome: Percentage of Patients With an ACR70 Response at Week 24, Based on ESR
Description: An ACR70 response is defined as having at least a 70% improvement in tender and swollen joints as well as a 70% improvement in 3 of 5 other criteria (patient assessment, physician assessment, pain scale, disability/functional questionnaire, and acute phase reactant value based on erythrocyte sedimentation rate [ESR]).
Time Frame: Baseline, 24 weeks
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Plus SOC | Belimumab 1 mg/kg Plus SOC | Belimumab 4 mg/kg Plus SOC | Belimumab 10 mg/kg Plus SOC
Number analyzed (Participants) | 69 | 72 | 71 | 71
percentage of participants | 2.9 | 5.6 | 1.4 | 2.8
Statistical Analysis 1: Comparison: Placebo Plus SOC vs Belimumab 1 mg/kg Plus SOC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4299, Likelihood ratio chi-squared — P-value was not adjusted for multiple testing; percent difference from placebo = 2.7, 95% CI 2-sided [-4.0 to 9.3]
Statistical Analysis 2: Comparison: Placebo Plus SOC vs Belimumab 4 mg/kg Plus SOC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5393, Likelihood ratio chi-squared — P-value was not adjusted for multiple testing; percent difference from placebo = -1.5, 95% CI 2-sided [-6.3 to 3.3]
Statistical Analysis 3: Comparison: Placebo Plus SOC vs Belimumab 10 mg/kg Plus SOC; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9769, Likelihood ratio chi-squared — P-value was not adjusted for multiple testing; percent difference from placebo = -0.1, 95% CI 2-sided [-5.6 to 5.4]

4. Secondary Outcome: Time to First ACR20 Response, Based on ESR
Description: The time to first ACR20 response (based on ESR) is defined as the time from the first dose to the first visit at which a patient first exhibited an ACR20 response, which may or may not have been sustained through Week 24.
Time Frame: 0 to 24 weeks
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo Plus SOC | Belimumab 1 mg/kg Plus SOC | Belimumab 4 mg/kg Plus SOC | Belimumab 10 mg/kg Plus SOC
Number analyzed (Participants) | 69 | 72 | 71 | 71
days | 112 [84 to NA] — 75th percentile could not be estimated because ≥40% of patients had no response | 109 [60 to 168] | 112 [49 to NA] — 75th percentile could not be estimated because ≥40% of patients had no response | 111 [57 to NA] — 75th percentile could not be estimated because ≥40% of patients had no response
Statistical Analysis 1: Comparison: Placebo Plus SOC vs Belimumab 1 mg/kg Plus SOC; Patients who required rescue RA medications were declared nonresponders, as were patients who dropped out or were missing Week 24 data. Patients who did not have any ACR response were censored at the last visit or exit visit, whichever occurred first. Patients who did not have an ACR response and discontinued from the study prior to study completion were censored at the last date on study; Test type: Superiority or Other; p = 0.1752, Log Rank — P-value was not adjusted for multiple testing
Statistical Analysis 2: Comparison: Placebo Plus SOC vs Belimumab 4 mg/kg Plus SOC; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.3440, Log Rank — P-value was not adjusted for multiple testing
Statistical Analysis 3: Comparison: Placebo Plus SOC vs Belimumab 10 mg/kg Plus SOC; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.4308, Log Rank — P-value was not adjusted for multiple testing

5. Secondary Outcome: Time to First ACR50 Response, Based on ESR
Description: Measure not posted because time to ACR50 response was unable to be determined due to the small number of patients achieving an ACR50 response in the study.
Time Frame: 0 to 24 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Time to First ACR70 Response, Based on ESR
Description: Measure not posted because time to ACR70 response was unable to be determined due to the small number of patients achieving an ACR70 response in the study.
Time Frame: 0 to 24 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Mean Change in Disease Activity Score 28 (DAS28) at Week 24
Description: DAS is a composite index of a patient's level of RA disease activity. DAS28 is an abbreviated version of DAS, using a subset of 28 joints in the assessment, calculated based on 4 variables: 1) number of tender joints out of a total of 28 joints, 2) number of swollen joints out of a total of 28 joints, 3) ESR, 4) patient's global assessment of disease activity based on a 100-mm visual analog scale. The calculation provides a number on a scale from 0 to 10 (>5.1=active disease; <3.2=well controlled disease; <2.6=remission). Change from baseline >1.2 = good response and ≤0.6 = non-response.
Time Frame: Baseline, 24 weeks
Population: Analysis was performed on a MITT population, defined as all patients who were randomized and received at least 1 dose of study agent and who had both a baseline and a Week 24 DAS28 score.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo Plus SOC | Belimumab 1 mg/kg Plus SOC | Belimumab 4 mg/kg Plus SOC | Belimumab 10 mg/kg Plus SOC
Number analyzed (Participants) | 69 | 72 | 71 | 70
scores on a scale | -0.9 (0.15) | -1.3 (0.18) | -0.9 (0.14) | -1.5 (0.15)
Statistical Analysis 1: Comparison: Placebo Plus SOC vs Belimumab 1 mg/kg Plus SOC; Missing data was handled by using last observation carried forward (LOCF) imputation; Test type: Superiority or Other; p = 0.0958, t-test, 2 sided — P-value was not adjusted for multiple testing
Statistical Analysis 2: Comparison: Placebo Plus SOC vs Belimumab 4 mg/kg Plus SOC; Missing data was handled by using LOCF imputation; Test type: Superiority or Other; p = 0.7864, t-test, 2 sided — P-value was not adjusted for multiple testing
Statistical Analysis 3: Comparison: Placebo Plus SOC vs Belimumab 10 mg/kg Plus SOC; Missing data was handled by using LOCF imputation; Test type: Superiority or Other; p = 0.0051, t-test, 2 sided — P-value was not adjusted for multiple testing

8. Secondary Outcome: Time to First DAS28 Response
Description: DAS28 response is defined as the time from the first dose to the first time at which a patient exhibited a "good" or a "moderate" improvement in RA disease activity, based on DAS28 improvements compared to baseline. Good response was defined as >1.2 change from baseline and DAS28 score ≤ 3.2. No response was defined as ≤ 0.6 change from baseline in DAS28 score or change between ≤ 1.2 and > 0.6 with a DAS28 score of > 5.1.
Time Frame: 0 to 24 weeks
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Arm/Group | Placebo Plus SOC | Belimumab 1 mg/kg Plus SOC | Belimumab 4 mg/kg Plus SOC | Belimumab 10 mg/kg Plus SOC
Number analyzed (Participants) | 69 | 72 | 71 | 71
days | 111 [56 to 168] | 82 [51 to 114] | 84 [33 to 168] | 57 [30 to 111]
Statistical Analysis 1: Comparison: Placebo Plus SOC vs Belimumab 1 mg/kg Plus SOC; Patients who required rescue RA medications were declared nonresponders, as were patients who dropped out or were missing Week 24 data. Patients who did not have good or moderate improvement in DAS28 were censored at the last visit or exit visit, whichever occurred first. Patients who did not have good or moderate improvement in DAS28 and discontinued from the study prior to study completion were censored at the last date on study; Test type: Superiority or Other; p = 0.0960, Log Rank — P-value was not adjusted for multiple testing
Statistical Analysis 2: Comparison: Placebo Plus SOC vs Belimumab 4 mg/kg Plus SOC; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.2859, Log Rank — P-value was not adjusted for multiple testing
Statistical Analysis 3: Comparison: Placebo Plus SOC vs Belimumab 10 mg/kg Plus SOC; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.0109, Log Rank — P-value was not adjusted for multiple testing

9. Secondary Outcome: Mean Change in Modified Total Sharp Score at Week 24
Description: The modified total Sharp score method was used to evaluate radiographs of hands/wrists for erosions (ERO) and joint space narrowing (JSN). The total modified Sharp score ranges from 0 (no radiographic damage) to 200 (worst possible radiographic damage) and is the sum of the normalized ERO score (range 0-100) and the normalized JSN score (range 0-100). Higher scores indicated more damage.
Time Frame: Baseline, 24 weeks
Population: Analysis was performed on a MITT population, defined as all patients who were randomized and received at least 1 dose of study agent and who had both a modified total Sharp score at baseline and at Week 24.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo Plus SOC | Belimumab 1 mg/kg Plus SOC | Belimumab 4 mg/kg Plus SOC | Belimumab 10 mg/kg Plus SOC
Number analyzed (Participants) | 67 | 70 | 66 | 68
scores on a scale | 0.7 (0.2) | 0.3 (0.2) | 0.3 (0.2) | 0.6 (0.2)
Statistical Analysis 1: Comparison: Placebo Plus SOC vs Belimumab 1 mg/kg Plus SOC; Missing data was handled by using LOCF imputation; Test type: Superiority or Other; p = 0.1940, t-test, 2 sided — P-value was not adjusted for multiple testing
Statistical Analysis 2: Comparison: Placebo Plus SOC vs Belimumab 4 mg/kg Plus SOC; Missing data was handled by using LOCF imputation; Test type: Superiority or Other; p = 0.2561, t-test, 2 sided — P-value was not adjusted for multiple testing
Statistical Analysis 3: Comparison: Placebo Plus SOC vs Belimumab 10 mg/kg Plus SOC; Missing data was handled by using LOCF imputation; Test type: Superiority or Other; p = 0.8707, t-test, 2 sided — P-value was not adjusted for multiple testing

10. Other Pre Specified Outcome: Adverse Events (AE) Overview
Description: Includes AEs reported in patients from the first dose of study agent throughout the study up to the Week 48/exit visit or 8 weeks following the last dose of study agent for patients who withdrew from this study or decided not to participate in the optional continuation protocol (LBRA99/NCT00583557).
Time Frame: Up to 56 weeks
Measure: Number; unit: percentage of participants
Groups:
- Open-label Extension Period: All Active: Includes all patients who completed the 24-week double-blind period and opted to continue in a 24-week open-label extension period. Belimumab patients received the same dose or were switched to 10 mg/kg at the investigator's discretion and former placebo patients received belimumab 10 mg/kg. AE onset may be during the extension phase or continuing from the double-blind period.
Arm/Group | Placebo Plus SOC | Belimumab 1 mg/kg Plus SOC | Belimumab 4 mg/kg Plus SOC | Belimumab 10 mg/kg Plus SOC | Open-label Extension Period: All Active
Number analyzed (Participants) | 69 | 72 | 71 | 71 | 237
percentage of participants
  Percent of patients with at least 1 AE | 89.9 | 84.7 | 90.1 | 93.0 | 91.6
  Percent of patients with at least 1 SAE | 7.2 | 6.9 | 7.0 | 8.5 | 11.0
  Percent of patients with an AE resulting in death | 1.5 | 0 | 0 | 1.4 | 0

ADVERSE EVENTS:
Time Frame: Up to 56 weeks
Description: Includes AEs reported in patients from the first dose of study agent throughout the study up to the Week 48/exit visit or 8 weeks following the last dose of study agent for patients who withdrew from this study or decided not to participate in the optional continuation protocol (LBRA99/NCT00583557).
Groups:
- Open-label Extension Period: All Active: Includes all patients who completed the 24-week double blind period and opted to continue in the 24-week open-label extension period. Belimumab patients received the same dose or were switched to 10 mg/kg at investigator discretion and former placebo patients received belimumab 10 mg/kg. AE onset may be during the extension phase or continuing from the double-blind period.
Arm/Group | Placebo Plus SOC | Belimumab 1 mg/kg Plus SOC | Belimumab 4 mg/kg Plus SOC | Belimumab 10 mg/kg Plus SOC | Open-label Extension Period: All Active
Serious Adverse Events (participants affected / at risk) | 5/69 | 5/72 | 5/71 | 6/71 | 26/237
Other Adverse Events (participants affected / at risk) | 50/69 | 47/72 | 48/71 | 54/71 | 165/237
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Plus SOC (N=69) | Belimumab 1 mg/kg Plus SOC (N=72) | Belimumab 4 mg/kg Plus SOC (N=71) | Belimumab 10 mg/kg Plus SOC (N=71) | Open-label Extension Period: All Active (N=237)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Spondylolisthesis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 2
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Clostridium colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Groin abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 | 1
Pneumonia primary atypical (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Medical device complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 3
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Intervertebral disc space narrowing (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Localised osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Obsessive-compulsive disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Cystocele (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Endometrial hypertrophy (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Plus SOC (N=69) | Belimumab 1 mg/kg Plus SOC (N=72) | Belimumab 4 mg/kg Plus SOC (N=71) | Belimumab 10 mg/kg Plus SOC (N=71) | Open-label Extension Period: All Active (N=237)
Diarrhoea (Gastrointestinal disorders) | 6 | 6 | 2 | 8 | 15
Mouth ulceration (Gastrointestinal disorders) | 2 | 1 | 4 | 0 | 3
Nausea (Gastrointestinal disorders) | 5 | 1 | 6 | 3 | 10
Fatigue (General disorders) | 4 | 5 | 6 | 7 | 18
Infusion site reaction (General disorders) | 1 | 4 | 0 | 2 | 4
Oedema peripheral (General disorders) | 4 | 3 | 9 | 3 | 25
Bronchitis (Infections and infestations) | 1 | 4 | 2 | 2 | 7
Nasopharyngitis (Infections and infestations) | 1 | 1 | 4 | 0 | 9
Sinusitis (Infections and infestations) | 2 | 3 | 7 | 3 | 13
Upper respiratory tract infection (Infections and infestations) | 9 | 6 | 9 | 10 | 38
Urinary tract infection (Infections and infestations) | 6 | 8 | 8 | 4 | 17
Contusion (Injury, poisoning and procedural complications) | 0 | 4 | 3 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 21 | 15 | 24 | 75
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2 | 2 | 18
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 | 4 | 6 | 11 | 21
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 6 | 4 | 4 | 14
Dizziness (Nervous system disorders) | 3 | 2 | 2 | 4 | 9
Headache (Nervous system disorders) | 4 | 7 | 5 | 8 | 12
Haematuria (Renal and urinary disorders) | 4 | 0 | 1 | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 8 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 7 | 1 | 2 | 7
Hypertension (Vascular disorders) | 2 | 4 | 2 | 2 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For multi-center trials, no investigator will be authorized to publish study results from an individual center until the multi-center trial results are published. All manuscripts and abstracts must be submitted to the sponsor for review at least 30 days prior to submission for publication or for presentation at a scientific meeting. Proposed abstracts and publications will be reviewed promptly.